CLINICAL TRIAL: NCT00444912
Title: A Pilot Cohort Study of AMD3100 in Combination With G-CSF and Rituximab Compared With AMD3100 in Combination With G-CSF Alone for Mobilization of BPCs in Patients With Relapsed or Refractory NHL or HD Prior to Autologous HPC Transplant
Brief Title: The Effect of Rituximab on Mobilization With AMD3100 (Plerixafor) Plus G-CSF in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma (NHL) or Hodgkin Disease (HD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMD31002113
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2010-07-29 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Non-Hodgkin Lymphoma; Hodgkin Disease
Keywords: AMD3100; stem cell mobilization; autologous transplant; Non-Hodgkin Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Granulocyte Colony-Stimulating Factor; plerixafor; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF plus plerixafor (Experimental): Participants with CD20- lymphoma
  Interventions: Drug: G-CSF plus plerixafor
- G-CSF plus plerixafor and rituximab (Experimental): Participants with CD20+ lymphoma
  Interventions: Drug: G-CSF plus plerixafor; Biological: rituximab

INTERVENTIONS:
Drug: G-CSF plus plerixafor — Participants underwent mobilization with G-CSF (7.5 µg/kg twice daily) for 4 days, administered by subcutaneous (sc) injection. On the evening of Day 4, participants received a dose of plerixafor (240 µg/kg), administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF (7.5 µg/kg) and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor. Participants were to continue to receive G-CSF twice daily and to receive the evening dose of plerixafor followed by apheresis the following morning for a maximum of 4 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Other Names: AMD3100; Mozobil
  Arms: G-CSF plus plerixafor
Drug: G-CSF plus plerixafor — Participants underwent mobilization with G-CSF (7.5 µg/kg twice daily) for 4 days, administered by subcutaneous (SC) injection. On the evening of Day 4, participants received a dose of plerixafor (240 µg/kg), administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF (7.5 µg/kg) and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor. Participants were to continue to receive G-CSF twice daily and to receive the evening dose of plerixafor followed by apheresis the following morning for a maximum of 4 aphereses or until ≥5*10^6 CD34+ cells/kg were collected.
  Other Names: Mozobil; AMD3100
  Arms: G-CSF plus plerixafor and rituximab
Biological: rituximab — Participants were given a weekly dose of rituximab 375mg/m2 by intravenous infusion for 1 week prior to and continuing until 2 weeks after the first dose of G-CSF.
  Other Names: Rituxan; MabThera
  Arms: G-CSF plus plerixafor and rituximab

SUMMARY:
Participants with non-Hodgkin lymphoma (NHL) or Hodgkin disease (HD) will be assigned to one of 2 arms based on the immunophenotype of their lymphoma.

(A)Participants with CD20(-) lymphoma will undergo mobilization with granulocyte colony-stimulating factor (G-CSF) and plerixafor.

(B) Participants with CD20(+) lymphomas will undergo mobilization with rituximab, G-CSF, and plerixafor. They will receive a weekly dose of rituximab beginning 1 week prior to, and continuing until 2 weeks after, the first dose of G-CSF.

Participants in both groups will receive G-CSF twice daily for 4 days. In the evening on Day 4, a dose of plerixafor will be administered. Apheresis will be initiated the next morning. Participants will continue to receive G-CSF twice daily and to receive the evening dose of plerixafor followed by apheresis the next morning for up to a total of 4 aphereses or until ≥5*10^6 CD34+ cells/kg are collected.

Participants who are transplanted will be monitored for the time to polymorphonuclear leukocytes (PMN), platelets (PLT), and lymphocyte engraftment. Follow-up assessments will be done at 100 days, and 6 and 12 months post-transplantation.

DETAILED DESCRIPTION:
This is a single-center, 2-arm, non-randomized, open-label study to evaluate the safety of plerixafor when used in combination with rituximab (Rituxan®) and granulocyte colony-stimulating factor (G-CSF) in patients with relapsed or refractory Hodgkin disease (HD) or non-Hodgkin lymphoma (NHL).

Participants will be assigned to one of 2 arms based on the immunophenotype of their lymphoma.

(A)Participants with CD20(-) lymphoma will undergo mobilization with G-CSF and plerixafor.

(B) Participants with CD20(+) lymphomas will undergo mobilization with rituximab, G-CSF, and plerixafor. They will receive a weekly dose of 375 mg/m2 rituximab by intravenous (iv) infusion beginning 1 week prior to, and continuing until 2 weeks after, the first dose of G-CSF.

Participants in both groups will receive 7.5 µg/kg G-CSF twice daily (morning and evening) for 4 days. In the evening (approximately 10:00 pm) on Day 4, a dose of plerixafor (240 µg/kg) will be administered. Apheresis will be initiated the next morning, approximately 10 to 11 hours after plerixafor is given. Participants will continue to receive G-CSF twice daily and to receive the evening dose of plerixafor followed by apheresis the next morning for up to a total of 4 aphereses or until ≥5*10^6 CD34+ cells/kg are collected.

Participants with an adequate number of autologous peripheral blood stem cells (PBSCs) collected by apheresis will be admitted to the study center for the administration of high-dose chemotherapy and autologous transplantation. After transplantation, the times to PMN, PLT, and lymphocyte engraftment will be measured. Participants will remain hospitalized until they achieve an absolute granulocyte count of >500/µl in the peripheral blood. Graft durability will be assessed at 100 days, and 6 and 12 months post-transplantation.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria (abbreviated list):

* Histological diagnosis of diffuse large cell lymphoma, B-cell, T-cell or anaplastic histologies; peripheral T-cell lymphoma; small non-cleaved Burkitt-like lymphoma; or Hodgkin disease. NOTE: Participants diagnosed at a facility outside of Emory University will have their diagnosis confirmed by Emory University pathologists prior to being enrolled in this study.
* Eligible for autologous transplantation.
* History of relapse of lymphoma following initial treatment with an anthracycline-containing regimen or disease that is refractory or progresses during initial therapy with an anthracycline-containing regimen.
* Immunophenotyping of the lymphoma at the time of diagnosis or relapse using flow cytometry or immunohistochemistry.
* Presence of clinically- and/or radiologically-documented, measurable, and/or evaluable disease at the time of relapse.
* Received 2 cycles of salvage chemotherapy.
* Complete response (i.e., normal physical examination, lymph nodes, lymph node masses, and bone marrow) or a partial response (i.e., decrease of ≧50% in the size of lymph nodes or lymph node masses or decrease in size of liver/spleen on physical exam) to at least one cycle of a salvage chemotherapy regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Absolute granulocytes count ≧1.0*10^9/l.
* Platelet count ≧75*10^9/l.
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) ≦2.5 times the upper limit of normal (ULN) or ≦5 times the ULN if liver involvement with lymphoma.
* Life expectancy of at least 3 months.
* >4 weeks since last cycle of chemotherapy.
* Patient has recovered from all acute toxic effects of prior chemotherapy.
* Signed informed consent.

Exclusion Criteria (abbreviated list):

* A second active malignancy (other than basal cell carcinoma of the skin).
* Uncontrolled central nervous system involvement by lymphoma.
* Positive/history of retroviral infection (HIV, HTLV-1).
* Active infection requiring antibiotics during planned lymphoma-related therapy.
* Previous treatment with high-dose chemotherapy or cytokine mobilization and hematopoietic progenitor cell transplantation.
* Continued evidence by morphology and flow cytometry of bone marrow involvement after at least one cycle of salvage chemotherapy.
* ≥3 cycles of salvage chemotherapy following documentation of lymphoma relapse or disease progression.
* (In patients with CD20(+) lymphoma) History of severe hypersensitivity reactions to rituximab.
* Positive pregnancy test in female patients.
* Lactating female patients.
* Previously received experimental therapy within 4 weeks of enrolling in this protocol or currently enrolled in another experimental protocol during G-CSF Mobilization Phase.
* Creatinine >1.5 times the ULN.
* Bilirubin >1.5 times the ULN.
* Ejection fraction <45%.
* Diffusion capacity of the lung for carbon monoxide (DLCO) <50%.
* Patients of childbearing potential unwilling to implement adequate birth control.
* A co-morbid condition that renders the patient at high risk from treatment complications.
* Residual acute medical condition resulting from prior chemotherapy.
* Documented history of ventricular arrhythmias during the last 3 years.
* Fever (temperature >38 °C/100.4 °F).
* Actual body weight exceeds 175% of ideal body weight.
* Participants who have deterioration of their clinical status or laboratory parameters between the time of enrolment and transplant (such that they no longer meet entry criteria) may be removed from study at the discretion of the treating physician, principal investigator, or sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- G-CSF and Plerixafor: Participants with CD20- lymphoma received granulocyte colony-stimulating factor (G-CSF) and plerixafor
- G-CSF and Plerixafor + Rituximab: Participants with CD20+ lymphoma received rituximab, G-CSF, and plerixafor
Period: Overall Study
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Started | 15 | 15
Received Plerixafor | 15 | 15
Received Transplant | 14 | 14
Completed | 12 | 13
Not Completed | 3 | 2
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant Failed Mobilization | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (11.3) | 46.5 (14.9) | 42.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 9 | 12 | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 12 | 10 | 22
  African-American | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Hispanic/Latino | 0 | 2 | 2
  Other | 0 | 2 | 2
Disease Diagnosis [Number; unit: Participants]
  Hodgkin disease (HD) | 14 | 4 | 18
  Non-Hodgkin lymphoma (NHL) | 1 | 11 | 12

OUTCOME MEASURES:

1. Primary Outcome: Summary of Adverse Events (AEs)
Description: Number of participants with adverse events (AEs) collected from Day 1 (start of G-CSF mobilization in participants with CD20- lymphoma or start of rituximab in participants with CD20+ lymphoma) to the day before starting chemotherapy. AEs were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for seriousness and relatedness to study treatment.
Time Frame: Day 1 and up to Day 59 (maximum time before start of chemotherapy)
Population: Safety Population: all participants who received at least 1 dose of study drug (G-CSF, plerixafor, or rituximab)
Measure: Number; unit: participants
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 15 | 15
participants
  Participants Reporting at Least 1 AE | 9 | 13
  Participant Count of Mild AEs | 7 | 12
  Participant Count of Moderate AEs | 2 | 0
  Participant Count of Severe AEs | 0 | 0
  Participant Count of Life-Threatening AEs | 0 | 1
  AEs by Relationship - Not Related | 1 | 0
  AEs by Relationship - Probably Not Related | 3 | 4
  AEs by Relationship - Possibly Related | 0 | 5
  AEs by Relationship - Probably Related | 2 | 3
  AEs by Relationship - Definitely Related | 3 | 1

2. Secondary Outcome: Median Cumulative Number of CD34+ Cells Collected During Apheresis
Description: Median total number of CD34+ cells collected during apheresis.
Time Frame: Days 5-8
Population: Full Analysis Set (FAS) includes all participants who received at least 1 dose of plerixafor.
Measure: Median (Full Range); unit: CD34+ cells (*10^6 / kg)
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 15 | 15
CD34+ cells (*10^6 / kg) | 7.4 [0.9 to 14.1] | 6.4 [2.5 to 10.9]

3. Secondary Outcome: Median Fold Increase in the Number of CD34+ Cells After Plerixafor Administration
Description: Fold Increase = (Pre-Apheresis CD34+ cells/Pre-Plerixafor CD34+ cells).
Time Frame: Days 4-5
Population: Evaluable population of participants with peripheral blood CD34+ measurements on Days 4 and 5.
Measure: Median (Full Range); unit: fold increase
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 6 | 11
fold increase | 2.4 [1.6 to 1321.3] | 2.5 [1.6 to 68.5]

4. Secondary Outcome: Median Number of Apheresis Days Required to Reach a Minimum of 3*10^6 CD34+ Cells/kg
Description: Median number of apheresis days in each treatment arm to collect a minimum of 3*10^6 CD34+ cells/kg.
Time Frame: Days 5-8
Population: Evaluable population of participants who achieved ≥3*10^cells/kg collected during apheresis.
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 14 | 14
days | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]

5. Secondary Outcome: Median Number of Apheresis Days Required to Reach the Target of 5*10^6 CD34+ Cells/kg
Description: Median number of apheresis days in each treatment arm to reach the target of 5*10^6 CD34+ cells/kg.
Time Frame: Days 5-8
Population: Evaluable population of participants who achieved ≥5*10^cells/kg collected during apheresis.
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 10 | 12
days | 1.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]

6. Secondary Outcome: Median Number of Days to Polymorphonuclear Leukocyte (PMN) Engraftment
Description: Median number of days from transplantation to PMN engraftment which was defined as PMN counts ≥0.5*10^9/L for 3 consecutive days or ≥1.0*10^9/L for 1 day. Time to engraftment corresponded to the first day that the criteria were met.
Time Frame: Days post transplantation (approximately Day 40)
Population: Evaluable population of participants who received a stem cell transplant and had PMN engraftment
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 14 | 14
days | 13.0 [11.0 to 21.0] | 13.5 [11.0 to 16.0]

7. Secondary Outcome: Median Number of Days to Platelet (PLT) Engraftment
Description: Median number of days from transplantation to PLT engraftment which was defined as platelet counts ≥20*10^9/L without transfusion for the preceding 7 days or platelet counts ≥50*10^9/L for one day. Time to engraftment corresponded to the first day that the criteria were met.
Time Frame: Days post transplantation (approximately Day 40)
Population: Evaluable population of participants who received a stem cell transplant and had PLT engraftment.
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 14 | 13
days | 21.0 [13.0 to 31.0] | 22.0 [16.0 to 28.0]

8. Secondary Outcome: Median Number of Days to Lymphocyte Engraftment
Description: Median number of days from transplantation to lymphocyte engraftment which was defined as lymphocyte counts ≥5*10^8/L. Time to engraftment corresponded to the first day that criteria were met.
Time Frame: Days post transplantation (approximately Day 40)
Population: Evaluable population of participants who received a stem cell transplant and had lymphocyte engraftment.
Measure: Median (Full Range); unit: days
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 14 | 14
days | 14.5 [9.0 to 32.0] | 14.0 [7.0 to 22.0]

9. Secondary Outcome: Median Level of CD19+CD2-CD14- B-cells Six Months Post-Transplant
Time Frame: Approximately 7 months (6 months post-transplant)
Population: Evaluable population of participants who received a stem cell transplant and had assessment performed 6 months post-transplant.
Measure: Median (Full Range); unit: cells / μL
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 5 | 4
cells / μL | 155.00 [61.00 to 311.00] | 0.50 [0.00 to 4.00]

10. Secondary Outcome: Median Level of CD19+CD2-CD14- B-cells Twelve Months Post-Transplant
Time Frame: 13 months (12 months post-transplant)
Population: Evaluable population of participants who received a stem cell transplant and had assessment performed 12 months post-transplant.
Measure: Median (Full Range); unit: cells / μL
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 6 | 6
cells / μL | 322.50 [189.00 to 518.00] | 236.00 [0.00 to 457.00]

11. Secondary Outcome: The Percentage of CD19+CD3-CD14- B-cells of the Total Cells on the First Apheresis Day
Time Frame: Day 5
Population: Full Analysis Set (FAS) includes all participants who received at least 1 dose of plerixafor.
Measure: Median (Full Range); unit: percentage of total cells
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 15 | 15
percentage of total cells | 2.83 [0.07 to 7.86] | 0.09 [0.01 to 0.39]

12. Secondary Outcome: Number of Participants With Durable Engraftment 12 Months After Transplantation
Description: The number of participants maintaining a durable graft 12 months after autologous transplantation. A durable graft is defined as the maintenance of normal blood counts.
Time Frame: Approximately 13 months (12 months post-transplant )
Population: Evaluable population of participants who received a stem cell transplant and had a 12-month assessment.
Measure: Number; unit: participants
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Number analyzed (Participants) | 14 | 14
participants | 12 | 13

ADVERSE EVENTS:
Time Frame: First day of G-CSF mobilization to the day prior to chemotherapy/ablative treatment in preparation for the first transplant. This timeframe includes G-CSF and plerixafor administration (rituximab if applicable), and the rest period.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
  Each AE table includes all events, regardless of reported relationship to study treatment or grade.
Arm/Group | G-CSF and Plerixafor | G-CSF and Plerixafor + Rituximab
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 9/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF and Plerixafor (N=15) | G-CSF and Plerixafor + Rituximab (N=15)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-CSF and Plerixafor (N=15) | G-CSF and Plerixafor + Rituximab (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Paraesthesia oral (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Catheter site discharge (General disorders) | 1 | 0
Catheter site erythema (General disorders) | 0 | 1
Catheter site pain (General disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Injection site erythema (General disorders) | 3 | 1
Injection site irritation (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 1
Injection site paraesthesia (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Urine pH increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.